CLINICAL TRIAL: NCT06056232
Title: Exploring the Mechanism of Mindfulness Intervention: Manipulating Distress the Dose of Tolerance Intervention Dose
Brief Title: Mechanisms of Mindfulness Intervention: Distress Tolerance Dose Manipulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E20230919
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Emotional Distress; Emotional Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIED group (Experimental): Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge, and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression, and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-normal version
- MIED+DT group (Experimental): The increase in distress tolerance dosage involves incorporating additional psychoeducational content related to distress tolerance and corresponding exercises to enhance distress tolerance within the MIED (Mindfulness Intervention for Emotional Distress) program.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-increase distress tolerance
- MIED-DT group (Experimental): The decrease in distress tolerance dosage entails reducing exercises related to distress tolerance within the MIED, such as interoceptive exposure exercises and challenging tasks.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-decrease distress tolerance

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-normal version — Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: MIED group
Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-increase distress tolerance — Increase the intervention dose of distress tolerance in Mindfulness Intervention for Emotional Distress (MIED). For example, including more emotion exposure tasks, materials from Facing Your Feelings.
  Arms: MIED+DT group
Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-decrease distress tolerance — Decrease the intervention dose of distress tolerance in Mindfulness Intervention for Emotional Distress (MIED). For example, including less emotion exposure tasks and interoceptive exposure tasks.
  Arms: MIED-DT group

SUMMARY:
This study hopes to:

1. explore whether an increase in the dosage of distress tolerance intervention corresponds to greater effectiveness of mindfulness intervention in alleviating emotional distress.
2. explore whether distress tolerance mediates the effects of mindfulness intervention on alleviating emotional distress.

DETAILED DESCRIPTION:
Epidemiological findings in "The Lancet Psychiatry" indicated that anxiety disorders, including generalized anxiety disorder, panic disorder, and social anxiety disorder, are the most prevalent category of disorders in China, with a lifetime prevalence of 7.6%. Depression follows closely with a lifetime prevalence of 6.8%. With the outbreak of the COVID-19 pandemic in 2020, the prevalence of both anxiety and depressive disorders increased. However, the current availability of psychological intervention resources in China is inadequate to meet the demand. This underscores the critical importance of developing effective and efficient psychological intervention approaches, as well as investigating their effectiveness and mechanisms to optimize intervention strategies.

In recent years, mindfulness-based interventions (MBIs) have been increasingly applied to alleviate emotional distress in both clinical and non-clinical populations, with their efficacy widely supported. Additionally, numerous researchers have explored the mechanisms underlying mindfulness and MBIs, proposing various theories. One of the mechanisms frequently suggested by researchers is exposure. However, there has been limited direct investigation into the mechanisms of exposure and its related processes or abilities. Distress tolerance (DT) is closely associated with exposure and is considered a common etiological factor or transdiagnostic characteristic of emotional distress, including anxiety and depression. Nevertheless, few studies have explored the mechanisms of how mindfulness interventions alleviate emotional distress from the perspective of exposure and the transdiagnostic characteristics of anxiety and depression. This lack of research hampers our ability to obtain sufficient information to develop or enhance mindfulness-based intervention methods to assist individuals with emotional disorders or highly emotionally distressed subclinical populations.

This study is grounded in the critical role of DT in the generation and maintenance of emotional distress, as well as the mindfulness principle of approaching pain with awareness and acceptance (non-judgmental and non-reactive). It posits that DT might be a potential mechanism through which mindfulness interventions alleviate emotional distress. Following the criteria for establishing mechanisms, this research investigates this issue. Based on the current state of research, DT as a mechanism for MBIs to alleviate emotional distress meets the plausibility criterion and partially satisfies the strong association criterion and experimental manipulation criterion. However, further research is needed to assess its consistency criterion, temporal precedence criterion, and gradient criterion.

The current study primarily focuses on the experimental manipulation and gradient criteria. The aim is to examine whether the mechanism of DT meets the experimental manipulation and gradient criteria by adjusting the content of the mindfulness intervention for emotional distress (MIED) program, which can directly impact distress tolerance and manipulate the dosage of distress tolerance intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.
* If taking medication, haven't changed for at least 4 weeks before intervention onset and no change in medicine is expected;
* Voluntary participation in this study and sign an informed consent form.

Exclusion Criteria:

* Subjects who have participated in mindfulness-based projects (especially MIED), and/or the current frequency of meditation practice is more than once a week;
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder, and generalized developmental disorder;
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-05 (Estimated); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Changes of Five Facet Mindfulness Questionnaire-short form during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Changes of Distress Tolerance Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Distress Tolerance Scale is used to measure Distress Tolerance. Scores range from 5 to 75, with higher scores indicating higher levels of Distress Tolerance.
Changes of Discomfort Intolerance Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Discomfort Intolerance Scale is used to measure Discomfort Intolerance. Scores range from 0 to 25, with higher scores indicating higher levels of discomfort intolerance.
Changes of Chinese Perceived Stress Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress.
Changes of 10-item Kessler Psychological Distress Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Changes of Overall Anxiety Severity and Impairment Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Changes of Overall Depression Severity and Impairment Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Changes of Beck Depression Inventory during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Beck Depression Inventory is a self-reported questionnaire measuring depression level.Scores range from 0 to 63, with higher scores indicating higher levels of depression.
Changes of Beck Anxiety Inventory during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Beck Anxiety Inventory is a self-reported questionnaire measuring Anxiety level.Scores range from 0 to 63, with higher scores indicating higher levels of Anxiety.
Changes of Athens Insomnia Scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.
Changes of Rumination during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  the Rumination subscale, extracted from the Rumination-Reflection Questionnaire, contains 12 items. Scores range from 5 to 60, with higher scores indicating higher levels of rumination.
Changes of Chinese version of the Brief Experiential Avoidance Questionnaire during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  Chinese version of the Brief Experiential Avoidance Questionnaire scale is used to measure experiential avoidance. Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Changes of Patient Health Questionnaire during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  he Patient Health Questionnaire is a self-reported questionnaire consisting of 18 items designed to measure the degree of being troubled by various common physical symptoms. Scores range from 0 to 30. 0~4 scores: no physical symptoms; 5~9 scores: mild physical symptoms; 10~14 scores: moderate physical symptoms; 15~30 scores: severe physical symptoms.
Changes of behavioral inhibition system/behavioral activation system (BIS/BAS) scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The BIS/BAS scale is a self-report questionnaire consisting of 18 items designed to assess the intensity of two motivational systems, namely the Behavioral Inhibition System (BIS) and the Behavioral Activation System (BAS). Scores on this scale can vary between 18 and 72, with elevated scores indicative of a greater tendency to avoid aversive outcomes and pursue goal-oriented outcomes.
Changes of Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) scale during the intervention | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  The Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) is a self-report questionnaire that aims to measure Interoceptive Awareness. Scores range from 0 to 165. Higher scores indicate higher ability or tendency in several domains including Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-regulation, Body Listening, and Trusting.

SECONDARY OUTCOMES:
The Paced Auditory Serial Addition Task-Computerized (PASAT-C) | at baseline (T0), at week 3(T1) and at week 5 (T2), at post-intervention (T3), and at 3 (T4) months follow-ups
  PASAT-C In this task, participants were presented with a series of numbers and were given the task of adding the last two numbers. They were given points for correct answers and unpleasant vocal feedback for incorrect answers. The task consists of four stages: (1) simple stage, which is the control condition of cognitive and motor function; (2) Latency test stage to determine the level of completion of the addition test; (3) distress induced stage, used to induce emotional pain; (4) distress tolerance stage, used to measure distress tolerance (i.e., the time before task termination).

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No